CLINICAL TRIAL: NCT00028743
Title: A Phase III Study of Cisplatin Plus Topotecan Followed by Paclitaxel Plus Carboplatin Versus Paclitaxel Plus Carboplatin as First Line Chemotherapy in Women With Newly Diagnosed Advanced Epithelial Ovarian Cancer
Brief Title: Combination Chemotherapy Regimens in Ovarian Epithelial Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Grupo Español de Investigación en Cáncer de Ovario (Other)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OV16; CAN-NCIC-OV16 (Other: PDQ); EORTC-55012 (Other: EORTC); GEICO-0101 (Other: GEICO); CDR0000069129 (Other: PDQ)
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cisplatin; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cisplatin, Topotecan, Paclitaxel plus Carboplatin (Active Comparator): Arm 1
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: paclitaxel; Drug: topotecan hydrochloride
- Paclitaxel plus Carboplatin (Active Comparator): Arm 2
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Arm 1 = 4 cycles vs Arm 2 = 8 cycles AUC5 (30 mins) day 1 of 21 day cycle
Drug: cisplatin — 4 cycles 50mg/m2 (60 mins) day 1 of 21 day cycle
  Arms: Cisplatin, Topotecan, Paclitaxel plus Carboplatin
Drug: paclitaxel — Arm 1 = 4 cycles vs Arm 2 = 8 cycles 175mg/m2 (3 hours) day 1 of 21 day cycle
Drug: topotecan hydrochloride — 4 cycles
  .75mg/m2 (30 mins) days 1-5 of 21 day cycle
  Arms: Cisplatin, Topotecan, Paclitaxel plus Carboplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving the drugs in different combinations may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating ovarian epithelial, primary peritoneal, or fallopian tube cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different combination chemotherapy regimens in treating patients who have stage IIB, stage III, or stage IV ovarian epithelial cancer , primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of cisplatin and topotecan followed by paclitaxel and carboplatin vs paclitaxel and carboplatin only, in terms of time to disease progression, in patients with newly diagnosed stage IIB-IV ovarian epithelial, primary peritoneal, or fallopian tube cancer.
* Compare the overall survival of patients treated with these regimens.
* Compare the clinical objective response rates in patients with measurable disease at baseline treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the CA 125 normalization rates in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, age (65 years and under vs over 65 years), and pre-randomization surgery (no debulking vs debulking with macroscopic residual disease less than 1 cm vs debulking with macroscopic residual disease 1 cm or greater vs debulking with no macroscopic residual disease). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive cisplatin IV over 60 minutes on day 1 and topotecan IV over 30 minutes on days 1-5 of courses 1-4 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 of courses 5-8.
* Arm II: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 of courses 1-8.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Planned interval debulking surgery should occur after course 3 or 4.

Quality of life is assessed at baseline; on day 1 of courses 3, 5, and 7; at the end of the last course; and at 3 and 6 months after study treatment completion.

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients (400 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIB-IV ovarian epithelial, primary peritoneal, or fallopian tube cancer

  * No borderline ovarian tumors
  * Residual disease allowed
* Fine needle aspiration showing an adenocarcinoma is allowed instead of open or true-cut biopsy if the following are true:

  * Presence of pelvic mass AND
  * Omental cake or other metastasis larger than 2 cm in the upper abdomen unless proven stage IV disease AND
  * Serum CA 125/carcinoembryonic antigen ratio at least 25 (if less than 25, a barium enema or colonoscopy and gastroscopy or radiological examination of the stomach should be negative for primary tumor within 6 weeks of study) AND
  * Normal mammography within 6 weeks of study

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than upper limit of normal

Cardiovascular:

* No clinically relevant atrial or ventricular arrhythmias
* No myocardial infarction (MI) within the past 6 months (pretreatment ECG as only evidence of MI allowed)
* No history of second- or third-degree heart blocks unless pacemaker implanted
* History of first-degree heart block allowed

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No complete bowel obstruction
* No prior allergic reaction to drugs containing Cremophor EL or compounds chemically related to study drugs
* No condition that would preclude high-volume saline diuresis
* No significant neurologic or psychiatric disorder that would preclude study compliance
* No active uncontrolled infection
* No neuropathy greater than grade 1
* No pre-existing hearing loss greater than grade 1
* No other concurrent serious illness or medical condition that would preclude study participation
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biological response modifiers or immunotherapy
* No concurrent prophylactic colony-stimulating factors (CSFs)

  * Concurrent therapeutic CSFs allowed

Chemotherapy:

* No prior chemotherapy for ovarian cancer
* No other concurrent cytotoxic agents

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* No prior radiotherapy for ovarian cancer

Surgery:

* No more than 6 weeks since prior planned pre-chemotherapy surgery for ovarian cancer
* Planned interval debulking allowed
* Concurrent second-look surgery allowed

Other:

* No prior non-surgical therapy for ovarian cancer
* No other concurrent investigational drug therapy
* No other concurrent anticancer treatment
* Concurrent enrollment on CAN-NCIC-OV13/EORTC 55971 allowed

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2001-08-31 (Actual); Primary Completion 2008-03-05 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Mar 2008

SECONDARY OUTCOMES:
Overall Survival | Dec 2012
Response Rates | March 2008
Toxic Effects | March 2008
Quality of Life | March 2008
CA125 Normalization Rates | March 2008

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Hoskins, MD, Study Chair — British Columbia Cancer Agency; Ignace B. Vergote, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (28):
- Canada (28):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - PEI Cancer Treatment Centre,Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoskins PJ, Vergote I, Stuart G, et al.: A phase III trial of cisplatin plus topotecan followed by paclitaxel plus carboplatin versus standard carboplatin plus paclitaxel as first-line chemotherapy in women with newly diagnosed advanced epithelial ovarian cancer (EOC) (OV.16). A Gynecologic Cancer Intergroup Study of the NCIC CTG, EORTC GCG, and GEICO. [Abstract] J Clin Oncol 26 (Suppl 15): A-LBA5505, 2008.